CLINICAL TRIAL: NCT03027193
Title: A Phase I Clinical Trial to Determine the Safety and Immunogenicity of the Candidate Mycobacterium Avium Subspecies Paratuberculosis (MAP) Vaccines ChAdOx2 HAV and MVA HAV in Healthy Adult Volunteers
Brief Title: A Study to Determine the Safety and Immunogenicity of a Candidate MAP Vaccines ChAdOx2 HAV and MVA in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HAV001
Record Dates: First submitted 2017-01-19; First posted 2017-01-23 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2019-05

CONDITIONS: Crohn Disease; Mycobacterium Avium Subspecies Paratuberculosis
Keywords: Vaccine; MAP
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1 (Experimental): Group 1 volunteers (n= 3 to 6) will be administered ChAdOx2 HAV, 5 x 10^9 vp through intramuscular route.
  Interventions: Biological: ChAdOx2 HAV
- Group 2 (Experimental): Group 2 volunteers (n= 3 to 6) will be administered ChAdOx2 HAV, 2.5 x 10^10 vp through intramuscular route.
  Interventions: Biological: ChAdOx2 HAV
- Group 3 (Experimental): Group 3 volunteers (n= 3 to 6) will be administered ChAdOx2 HAV, 5 x 10^10 vp through intramuscular route.
  Interventions: Biological: ChAdOx2 HAV
- Group 4 (Experimental): Group 4 volunteers (n= 3) will be administered MVA HAV, 5 x 10^7 pfu through intramuscular route.
  Interventions: Biological: MVA HAV
- Group 5 (Experimental): Group 5 volunteers (n= 3) will be administered MVA HAV, 2 x 10^8 pfu through intramuscular route.
  Interventions: Biological: MVA HAV
- Group 6 (Experimental): Group 6 volunteers (n= 10) will be administered ChAdOx2 HAV, 5 x 10^10 vp followed by MVA HAV, 2 x 10^8 pfu (8 weeks apart) through intramuscular route.
  Interventions: Biological: ChAdOx2 HAV; Biological: MVA HAV

INTERVENTIONS:
Biological: ChAdOx2 HAV — The ChAdOx2 HAV vaccine consists of the replication-deficient simian adenovirus vector ChAdOx2, containing the Mycobacterium avium subspecies paratuberculosis (MAP) antigens
  Arms: Group 1; Group 2; Group 3; Group 6
Biological: MVA HAV — The MVA HAV vaccine consists of the replication deficient modified vaccinia virus Ankara (MVA) containing the Mycobacterium avium subspecies paratuberculosis (MAP) antigens.
  Arms: Group 4; Group 5; Group 6

SUMMARY:
A phase I dose escalation study to assess the safety and immunogenicity of the candidate vaccines ChAdOx2 HAV and MVA HAV in healthy volunteers.

Volunteers will be recruited and vaccinated in Oxford, England.

All vaccinations will be administered intramuscularly. Three different doses of the ChAdOx2 HAV will be tested (5x10^9 vp, 2.5x10^10 vp and 5x10^10vp). MVA HAV will be assessed at 2 different doses (5x10^7 and 2x10^8 pfu)

The total duration of the study will be 52 weeks from the day of enrolment for volunteers receiving ChAdOx2 HAV only, 12 weeks for volunteers receiving MVA HAV only and 20 weeks for volunteers receiving ChAdOx2 HAV and MVA HAV.

DETAILED DESCRIPTION:
This is a phase I, open label, dose escalation trial to assess the safety and immunogenicity of the ChAdOx2 and MVA HAV vaccines against Mycobacterium avium subspecies paratuberculosis (MAP) in healthy volunteers

There will be 5 study groups with a total of 28 volunteers. ChAdOx2 HAV will be administered intramuscularly as a single vaccination at 3 different doses: 5x10^9 vp (group 1), 2.5x10^10 (group 2) and 5x10^10 vp (group 3) and as a prime vaccine in group 6 (prime/boost group). MVA HAV will be administered intramuscularly as a single vaccination at 2 different doses: 5x10^7 pfu (group 4), 2x10^8 pfu (group 5) and as a boost vaccine in group 6 (prime/boost group)

Vaccination of groups will be sequential from Group 1 to Group 6 with interim safety reviews prior to dose escalation

Volunteers will be recruited and undergo screening visits, vaccination and clinic visits post-vaccination at the trial site. Blood samples for safety and immunology purposes will be performed on the visit time points indicated in the schedule of attendances.

Safety will be assessed by the frequency, incidence and nature of adverse events and serious adverse events arising during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged 18 to 50 years
2. Able and willing (in the Investigator's opinion) to comply with all study requirements
3. Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner
4. For females only, willingness to practice continuous effective contraception (see below) during the study and a negative pregnancy test on the day(s) of screening and vaccination
5. Agreement to refrain from blood donation during the course of the study
6. Provide written informed consent

Exclusion Criteria:

1. Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the study period
2. Prior receipt of an investigational vaccine likely to impact on interpretation of the trial data.
3. Prior receipt of an adenoviral vectored vaccine in the last 12 months
4. Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
5. Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
6. History of allergic disease or reactions likely to be exacerbated by any component of the vaccine
7. Any history of hereditary angioedema, acquired angioedema, or idiopathic angioedema.
8. Any history of anaphylaxis in relation to vaccination
9. Pregnancy, lactation or willingness/intention to become pregnant during the study
10. History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
11. History of serious psychiatric condition likely to affect participation in the study
12. Bleeding disorder (eg. Factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venepuncture
13. Any other serious chronic illness requiring hospital specialist supervision
14. Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week
15. Suspected or known injecting drug abuse in the 5 years preceding enrolment
16. Seropositive for hepatitis C (antibodies to HCV)
17. Seropositive for hepatitis B surface antigen(HBsAg)
18. Any clinically significant abnormal finding on screening biochemistry or haematology blood tests or urinalysis
19. Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data
20. Inability of the study team to contact the volunteer's GP to confirm medical history and safety to participate.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-01-16 (Actual)

PRIMARY OUTCOMES:
Occurrence of solicited and unsolicited local and systemic adverse events | up to 28 days following vaccination
  The specific endpoints for safety and reactogenicity will be actively and passively collected data on adverse events. Change from baseline for safety laboratory measures will also be collected. Occurrence of serious adverse events will be collected during the whole study duration

SECONDARY OUTCOMES:
Measures of Immunogenicity of ChAdOx2 HAV and MVA HAV | Approximately 2 months post each vaccination
  To assess the immunogenicity of ChAdOx2 HAV and MVA HAV in healthy adult volunteers when administered alone and in a prime-boost regimen

CONTACTS AND LOCATIONS:
Overall Officials: Adrian V Hill, DPhill FRCP, Principal Investigator — Centre for Clinical Vaccinology and Tropical Medicine, Churchill Hosptal, Oxford, United Kingdom
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, Churchill Hospital, Oxford, United Kingdom